CLINICAL TRIAL: NCT06656364
Title: Esprit BTK Post-Approval Study (Esprit BTK PAS)
Brief Title: Esprit BTK Post-Approval Study
Acronym: EspritBTKPAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10519
Record Dates: First submitted 2024-10-15; First posted 2024-10-24 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-05

CONDITIONS: Chronic Limb-Threatening Ischemia
Keywords: ABT-CIP-10519; Esprit BTK System; Infrapopliteal lesions; Post-approval study
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Esprit BTK System (Experimental): This device, manufactured by Abbott Medical, is intended to be used for improving luminal diameter in infrapopliteal lesions in patients with CLTI.
  Interventions: Device: Esprit BTK System

INTERVENTIONS:
Device: Esprit BTK System — The Esprit BTK System is a resorbable polymeric scaffold with the everolimus drug and a resorbable polymeric coating mounted on a balloon dilatation catheter.

SUMMARY:
The Esprit BTK PAS is a prospective, single-arm, multi-center observational study to assess the continued safety and effectiveness of the Esprit™ BTK Everolimus Eluting Resorbable Scaffold System under commercial use, in patients with diseased infrapopliteal lesions causing CLTI (Chronic Limb-Threatening Ischemia) in a real-world setting. The clinical investigation will be conducted at up to 50 sites in the United States (US) and additional sites may be added outside of the US (OUS). Approximately 200 patients with a minimum of 50% of patients in the US will be registered in the clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria

  1. Subject must provide written informed consent prior to any study-specific procedures which are not considered standard of care at the site.

     1. Informed consent can be obtained up to 3 days post-procedure or prior to discharge whichever comes first.
     2. Subject, or a legally acceptable representative must provide written informed consent per site IRB/EC requirements.
  2. Subject must be at least 18 years of age.
  3. Subject has evidence of symptomatic Chronic Limb-Threatening Ischemia (CLTI) with infrapopliteal lesions.
* Anatomic Inclusion Criteria

  1. Subjects who have lesion(s) in an infrapopliteal vessel with reference vessel diameter ≥ 2.5 mm and ≤ 4.0 mm.
  2. Target lesion(s) must have ≥ 70% stenosis, per visual assessment at the time of the procedure. If needed, quantitative imaging (angiography and intravascular imaging) can be used to aid accurate sizing of the vessels.

Exclusion Criteria:

* General Exclusion Criteria

  1. Subjects who have contraindications to the Esprit BTK System per the instruction for use (IFU).
  2. Subject is currently participating in another clinical investigation.
  3. Subject is unable or unwilling to provide written consent prior to enrollment.
  4. Subject with life expectancy ≤ 1 year.
  5. Subject with an unsalvageable limb (as per physician assessment at the time of the index procedure), who is likely to get a below-the-knee amputation.
* Anatomic Exclusion Criteria

  1. Subject has in-stent restenosis in the target vessel or requires treatment with a metallic stent in the target vessel during the index procedure.
  2. Subject had been previously treated with Esprit BTK Scaffold(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Primary Effectivenes Endpoint(s): Freedom from clinically-driven target lesion revascularization (CD-TLR) | At 1 year
  This effectiveness endpoint was chosen because it allows to assess whether Esprit BTK is effective at maintaining patency (CD-TLR).
Primary Safety Endpoint(s):MALE at 6 months + POD at 30 days (Major Adverse Limb Event + Peri-Operative Death) | 6 months + 30 days
  This safety endpoint was chosen because it is a commonly used endpoint to assess the safety of devices used in lower limb treatment, including treatment of lesions below the knee. Additionally, this endpoint assesses whether the device is associated with acute and sub-acute harm such as death and limb loss.

SECONDARY OUTCOMES:
All-cause mortality | Discharge (between 0 and 10-days post-index procedure), 30 days, 90 days (only for subjects with index wound), 6 months, 1 year, 2 years, 3 years
Amputation (minor, major) | Discharge (between 0 and 10-days post-index procedure), 30 days, 90 days (only for subjects with index wound), 6 months, 1 year, 2 years, 3 years
Amputation-free survival | Discharge (between 0 and 10-days post-index procedure), 30 days, 90 days (only for subjects with index wound), 6 months, 1 year, 2 years, 3 years
Ankle-Brachial Index (ABI)/Toe-Brachial Index (TBI) progression over time | Discharge (between 0 and 10-days post-index procedure), 30 days, 90 days (only for subjects with index wound), 6 months, 1 year, 2 years, 3 years
Rutherford Becker category evolution over time | Discharge (between 0 and 10-days post-index procedure), 30 days, 90 days (only for subjects with index wound), 6 months, 1 year, 2 years, 3 years
Wound healing, as assessed by investigator | Discharge (between 0 and 10-days post-index procedure), 30 days, 90 days (only for subjects with index wound), 6 months, 1 year, 2 years, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ramon L Varcoe, MBBS, MS, FRACS, PHD, Principal Investigator — Prince of Wales Private Hospital, Randwick, NSW, Australia; Sahil Parikh, MD, Principal Investigator — New York Presbyterian Hospital, New York, NY; Brian G Derubertis, MD, Principal Investigator — New York Presbyterian/Cornell, New York, NY
Locations (35):
- United States (32):
  - HonorHealth, Scottsdale, Arizona
  - Pima Heart and Vascular Clinical Research, Tucson, Arizona
  - UCSF Fresno, Fresno, California
  - Good Samaritan Hospital, Los Angeles, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Ansaarie Cardiac and Endovascular Center of Excellence, Saint Augustine, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Grady Clinical Research Center, Atlanta, Georgia
  - Archbold Medical Center, Thomasville, Georgia
  - SIU School of Medicine, Springfield, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - Charlton Memorial Hospital, Fall River, Massachusetts
  - Jackson Heart Clinic, Jackson, Mississippi
  - North Mississippi Medical Center, Tupelo, Mississippi
  - New York University Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - New York Presbyterian Hospital-Cornell University, New York, New York
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Staten Island University Hospital - North, Staten Island, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - Ascension St. John Jane Phillips, Bartlesville, Oklahoma
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Johnson City Medical Center Hospital, Johnson City, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - Park Plaza Hospital, Houston, Texas
- Queen Mary Hospital, Hong Kong, HK SAR, Hong Kong
- Auckland City Hospital, Auckland, New Zealand
- Al Qassimi Hospital, Sharjah city, Emirate of Sharjah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No